CLINICAL TRIAL: NCT03720340
Title: The Open and Multi-center Phase III Clinical Study of Interleukin-11 in the Prevention and Treatment of Radioactive Oral Mucitis
Brief Title: Interleukin-11 Can Prevent and Treat of Radioactive Oral Mucitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen yuanyuan, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2018-180
Record Dates: First submitted 2018-10-10; First posted 2018-10-25 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Acute Radiation Oral Mucositis; Recombinant human interleukin-11; oral microflora
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Interleukin-11; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant human interleukin-11 (Active Comparator): Mixture of 1.5 mg recombinant human interleukin -11(IL-11) and 10ml 0.9% normal saline(NS) was administered twicely to patients through respiratory tract.
  Interventions: Drug: Recombinant Human Interleukin-11; Drug: Saline
- Saline (Placebo Comparator): Only 10ml 0.9% NS was administered twicely to patients through respiratory tract.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Recombinant Human Interleukin-11 — Recombinant Human Interleukin-11 was administed through respiratory tract.
  Arms: Recombinant human interleukin-11
Drug: Saline — saline was administed through respiratory tract

SUMMARY:
Radiation induced oral mucositis which may result in reduced quality of life is commonly seen during radiotherapy, especially combined with chemotherapy. This study is a prospective, multicenter, and exploratory study. The aim of this study is to explore predictive factors of acute radiotherapy induced oral mucositis in nasopharyngeal carcinoma patients treated with radio-chemotherapy and reduce incidence of oral mucositis by using recombinant human interleukin -11.

DETAILED DESCRIPTION:
All nasopharyngeal patients received radical treatment including neo-adjuvant chemotherapy and concurrent chemo-radiotherapy. Oral pharyngeal swabs and stool specimen were collected 3times:before neo-adjuvant chemotherapy,before concurrent chemo-radiotherapy and concurrent chemo-radiotherapy finishied. Patients were randomly divided into two groups randomly. IL-11 was used in experience group and control group, saline.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of nasopharyngeal carcinoma.
2. 8th version American Joint Committee on Cancer (AJCC) stage I-IVB.
3. Age must beetween 18-75.
4. Performance status must be 0 or 1 according to Eastern Cooperative Oncology Group.
5. Adequate bone marrow, renal, and hepatic function.

Exclusion Criteria:

1. chemotherapy with fluorouracil drugs; Allergies to recombinant human interleukin-11.
2. Treatment with palliative intent.;Previous malignancy.
3. Pregnancy or lactation.
4. A history of previous radiotherapy, chemotherapy, or surgery (except diagnostic) to the primary tumor or nodes.
5. Diabetes, oral mucositis and senile dry stomatitis.
6. Any severe coexisting disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe acute radioactive oral mucitis | through study completion, an average of 5mouth
  Radiation Therapy Oncology Group/European Organization for research and treatment acute radiation morbidity scoring criteria. Grade 0: No change over baseline, Grade 1: Injection/ may experience mild pain not requiring analgesic, Grade 2: Patchy mucositis which may produce an inflammatory serosanguinitis discharge/ may experience moderate pain requiring analgesia, Grade 3: Confluent fibrinous mucositis/ may include severe pain requiring narcotic, Grade 4: Ulceration, hemorrhage or necrosis, Grade 5: death (Higher score equals to worse outcome).

SECONDARY OUTCOMES:
Comparison of the occurrence time of severe acute radioactive oral mucitis in two groups | first day from radiation to the date 3 degree acute radioactive oral mucitis occurred
  RGOT/ CTCA
last period of severe acute radioactive oral mucitis | through study completion, an average of 5month
  RGOT/ CTCA
Changes in oral flora | through study completion, an average of 5month
  Changes in oral flora during treatments
Changes in intestinal flora | through study completion, an average of 5month
  Changes in oral intestinal during treatments
Nutritional status | through study completion, an average of 5month
  Nutrition Risk Screening NRS-2002 Assessment Comparison of Nutritional Status of Two Groups of Patients
Comparison of quality of life | through study completion, an average of 5month
  Life Quality Measurement Scale H&N35 Comparison of quality of life between two groups of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No